CLINICAL TRIAL: NCT06561516
Title: Effects of Red Ginseng on Gastrointestinal Symptoms and Microbiota After Surgery for Gastrointestinal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, In Gyu Kwon, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2022-0046
Record Dates: First submitted 2024-08-04; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Stomach Cancer; Pancreatobiliary Cancer; Colorectal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Colorectal Neoplasms | interventions — Asian ginseng

STUDY DESIGN:
Intervention Model Description: We randomly assign enrolled patients in two groups, Red ginseng group and Control group. The Red ginseng group will consume red ginseng (ginsenoside 500mg/T) for three months starting one month after surgery. Microbiome analysis will be conducted before surgery and at four months after surgery to investigate the prebiotic effects of red ginseng on gut microbiota distribution. The control group will not recieve any intervention during the experimental periods.
Who Masked: Investigator
Masking Description: The participating physicians in the study are kept unaware of which group each patient belongs to. However, patients are randomly divided into the Red ginseng and Control groups by research nurses, and they become aware of their group assignment (whether they will take red ginseng tablets or not) in a single-blind study format.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red ginseng group (Experimental): The Red ginseng group will consume red ginseng (ginsenoside 500mg/T) for three months starting one month after surgery. Patients take 2 tablets of 500mg ginsenoside twice daily.
  Interventions: Procedure: Arm I (Red ginseng)
- Control group (No Intervention): The control group will not receive any intervention during the experimental periods.

INTERVENTIONS:
Procedure: Arm I (Red ginseng) — Step 1. Confrim the inclusion and exclusion criteria to select participants and abtain informed consent before surgery.
  Step 2. Before surgery, research nurses randomly assign patients to either the Red ginseng or Control group (single-blind study).
  Step 3. Blood tests and stool samples following rectal enema are collected from all patients before surgery.
  Step 4. Depending on the type of gastrointestinal cancer (stomach cancer, pancreatobiliary cancer, colorectal cancer), radical resection surgery is performed.
  Step 5. From 1 to 4 months after surgery, a three months period is designated for the Red ginseng group to take red ginseng tablets as instructed, with compliance assessements included.
  Step 6. Four months after surgery, blood tests and stool samples are collected from all patients.
  Step 7. After obtaining samples from the final registered patients, we will commission a contracted institution to conduct microbiome analysis test.
  Arms: Red ginseng group

SUMMARY:
After surgery for gastrointestinal cancer (stomach cancer, pancreaticobiliary cancer, colorectal cancer), many patients experiences various symptoms such as weight loss, diarrhea, constipation and excessive gas due to structural and functional changes in the gastrointestinal tract. These changes are thought to be influenced by alterations in gut microbiota following surgery, but prospective studies are still lacking. It is anticipated that the prebiotic effects of red ginseng may lead to positive changes in total gut bactera after gastrointestinal caner surgery.

Through this study, Investigators aim to investigate the impact of red ginseng consumption on gut microbiota composition, gastrointestinal symptoms, and nutritional status improvement following surgery for gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed with gastrointestinal cancers (stomach cancer, pancreatobiliary cancer, colorectal cancer) prior to surgery.
2. Clinically staged and anticipated to not receive adjuvant chemotherapy after surgery.
3. Eligible for complete surgical resection (R0 resection).
4. ASA (American Society of Anesthesiologists) score of 3 or below.
5. Intereseted in health functional foods.
6. Not consumed probiotics or prebiotics for at least three months prior to study enrollment.
7. Willing to refrain from consuming additional probiotics or prebiotics during the study period, apart from the provided red ginseng tablets.

Exclusion Criteria:

1. Patients aged 80 years or older.
2. Patients who received neoadjuvant therapy before surgery.
3. Patients with underlying gastrointestinal disorders (e.g., inflammatory bowel disease, ulcerative colitis, Crohn's disease, galactose intolerance, lactase deficiency, glucose-galactose malabsorption, short bowel syndrome, other hereditary gastrointestinal diseases, and autoimmune diseases).
4. Patients unable to orally consume red ginseng tablets.
5. Patients with a history of previous abdominal organ surgery, radiation therapy, or chemotherapy.
6. Patients with intestinal obstruction before surgery.
7. Patients regularly taking probiotic or prebiotic supplements.
8. Patients requiring formation of an ileostomy after surgery.
9. Patients with uncontrolled diabetes that may affect gastrointestinal function.
10. Patients with underlying conditions such as liver failure or renal failure.
11. Patients allergic to red ginseng.
12. Patients who received more than two weeks of antibiotic treatment during hospitalization.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Changes in microbiome composition based on the consumption or non-consumption of red ginseng following gastrointestinal cancer surgery. | 4 months after surgery
  We observe changes in total gut bacteria following gastrointestinal cancer surgery based on the consumption of red ginseng through analysis of fecal microbiome.

SECONDARY OUTCOMES:
Improvement of gastrotintestinal symptoms | 4 months after surgery
  EORTC QLQ-30 questionaire: gas expulsion level and discomfort caused by gas expulsion)
Improvement of bowel habits | 4 months after surgery
  Bowel habit questionnaire
Nutritional Indicators | 4 months after surgery
  Blood test- lymphocyte counts
Nutritional Indicators | 4 months after surgery
  Blood test- albumin level
Nutritional Indicator | 4 months after surgery
  Blood test- total protein level

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severacne Hospital Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No